CLINICAL TRIAL: NCT00005002
Title: A Randomized, Double-Blind, Adjuvant-Controlled, Multicenter Study to Compare the Virologic and Immunologic Effect of Highly Active Antiretroviral Therapy (HAART) Plus Remune Versus HAART Plus Incomplete Freund's Adjuvant (IFA) in Antiretroviral-Naive Patients Infected With Human Immunodeficiency Virus Type 1 (HIV-1)
Brief Title: Effectiveness of Treating HIV-Positive Patients With an HIV Vaccine (Remune)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: B009; AG1661-202
Record Dates: First submitted 2000-03-21; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-08

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; CD4 Lymphocyte Count; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; remune; Combivir
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination; HIV-1 immunogen, incomplete Freund's adjuvant; Nelfinavir

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Biological: HIV-1 Immunogen
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to see if it is effective to add an HIV vaccine (Remune) to the anti-HIV drug combination of Combivir (zidovudine plus lamivudine) and nelfinavir.

DETAILED DESCRIPTION:
All patients begin HAART at study entry (Day 1). Patients with a plasma HIV-1 RNA level less than or equal to 2,000 copies/ml at Week 8 are randomized to receive Remune or Incomplete Freund's Adjuvant (IFA) at Week 9. Patients who do not achieve a plasma HIV-1 RNA level of less than or equal to 2,000 copies/ml at Week 8 are not randomized and are terminated from the study. These patients are eligible to receive funding for up to a 3-month supply of nelfinavir (Viracept) and Combivir. Randomized patients receive Remune or IFA at Week 9 and approximately every 12 weeks thereafter until study completion (when the last patient reaches Week 48). Patients are considered virologic failures if they (1) fail to achieve a virologic response by Week 48 or (2) after achieving a virologic response, have a virologic relapse. Regardless of their previous response status, patients whose plasma HIV-1 RNA level increases to greater than 2,000 copies/ml while they are receiving protocol-specified HAART are eligible to receive salvage therapy and continue to receive Remune or IFA until study completion. Study visits occur at screening, Day 1, Weeks 4, 8, 9, 12, and then every 4 weeks thereafter until the last patient reaches Week 48. Patients who complete this study are eligible to participate in a rollover study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 13 years old (consent of parent or guardian required if under 18).
* Have a viral load of at least 10,000 copies/ml.
* Have a CD4 count of at least 250 cells/mm3.
* Have never taken any anti-HIV drugs before.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 688

CONTACTS AND LOCATIONS:
Locations (1):
- Agouron Pharmaceuticals Inc, San Diego, California, United States